CLINICAL TRIAL: NCT01815515
Title: Evaluation of 18F-DCFBC PSMA-based PET Imaging for Detection of Metastatic Prostate Cancer.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J12113; NA_00052383 (Other: JHM IRB)
Record Dates: First submitted 2013-03-18; First posted 2013-03-21 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — N-(N-((S)-1,3-Dicarboxypropyl)carbamoyl)-4-(18F)fluorobenzyl-L-cysteine

ARMS (1):
- 18F-DCFBC (Experimental): Participants with hormone-naive prostate cancer (HNPC) and castration-resistant prostate cancer (CRPC) with metastatic lesions detected on conventional imaging modalities (contrast-enhanced computed tomography [CECT] and bone scintigraphy [BS]) undergo PET imaging with 18F-DCFBC radiotracer.
  Interventions: Drug: 18F-DCFBC

INTERVENTIONS:
Drug: 18F-DCFBC — 18F-DCFBC is a radiofluorinated small-molecule inhibitor of prostate-specific membrane antigen (PSMA).
  A bolus of 10 mCi (370 MBq) [9-11 mCi (333-407 MBq)] of 18F-DCFBC will be injected into the IV line by slow IV push.
  Other Names: N-[N-[(S)-1,3-dicarboxypropyl]carbamoyl]-4-18F-fluorobenzyl-L-cysteine

SUMMARY:
This research is being done to see if an investigational radioactive drug called 18F-DCFBC can help us find cancer that has spread (metastatic disease) from its original site in people who have cancer in their prostate to other parts of their body.

DETAILED DESCRIPTION:
The objective of this study is to evaluate a radiolabeled urea-based small molecule inhibitor of prostate-specific membrane antigen (PSMA), [18F]DCFBC (DCFBC) PET imaging for detection of metastatic prostate cancer. PSMA is a well characterized histological marker of prostate cancer tumor aggressiveness and metastatic potential. The investigators propose to assess the ability of DCFBC PET to detect metastatic prostate cancer by visual qualitative and quantitative SUV analysis. Correlation will be made to sites of suspected metastatic disease detected by standard conventional imaging modalities (CIM) for prostate cancer which includes IV contrast CT of chest/abdomen/pelvis and whole body bone scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of prostate cancer
2. Radiologic evidence of new or progressive metastatic disease demonstrated on anatomical imaging (CT, MRI, or ultrasound), bone scintigraphy, [18F]Sodium Fluoride PET, and/or [18F]FDG PET
3. Rising PSA on two observations taken at least 1 week apart
4. Adequate peripheral venous access or available central venous catheter access for radiopharmaceutical administration
5. Patient can remain on androgen deprivation therapy if on the same regimen prior to documentation of progressive metastatic disease
6. Patient cannot start a new therapy for prostate cancer prior to study radiopharmaceutical imaging
7. Patient is judged by the Investigator to have the initiative and means to be compliant with the protocol and be within geographical proximity to make the required study visits
8. Patients or their legal representatives must have the ability to read, understand and provide written informed consent for the initiation of any study related procedures

Exclusion Criteria:

1. Patient has been treated with an investigational drug, investigational biologic, or investigational therapeutic device within 14 days prior to study radiotracer administration
2. Prior radiation therapy, chemotherapy, or androgen-deprivation therapy within 2 weeks prior to study radiotracer administration (Washout is one half-life of the drug or 2 weeks, whichever is longest)
3. Initiation of new therapy for progressive metastatic disease since radiographic documentation of progression.
4. Serum creatinine > 3 times the upper limit of normal
5. Total bilirubin > 3 times the upper limit of normal
6. Liver Transaminases > 5times the upper limit of normal
7. Unable to lie flat during or tolerate PET/CT
8. Prior history of any other malignancy within the last 2 years, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Szabo, M.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 participants enrolled, 5 screen failures, therefore only 17 participants started the study.
Period: Overall Study
Arm/Group | 18F-DCFBC
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18F-DCFBC
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (7.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
Prostate specific antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 95.6 (141.26)
Serum folate [Count of Participants; unit: Participants]
  Normal range (2.5-20 ng/mL) | 11
  21-24 ng/mL | 1
  High (>24 ng/mL) | 5
Red cell folate [Mean (Full Range); unit: ng/mL] — Normal range = 160-855 ng/mL Population: Data was not available in 4 participants
  ng/mL
    number analyzed (Participants) | 13
    (all) | 550.69 [268 to 1049]
Testosterone <20 ng/mL [Count of Participants; unit: Participants] | 8
Testosterone [Mean (Full Range); unit: ng/mL] — Population: Mean testosterone level (ng/mL) for participants with values other than "<20 ng/mL"
  ng/mL
    number analyzed (Participants) | 9
    (all) | 396.33 [245 to 746]
Prior prostate cancer therapy [Count of Participants; unit: Participants]
  Prostatectomy | 7
  Androgen deprivation | 8
  Docetaxel | 2
  Tasquinimod | 1
  Abiraterone | 1
  External-beam radiation to the pelvis | 7
  External-beam radiation to the right hip | 1
  External-beam radiation to the spine | 1
  Prostate brachytherapy | 1
  Radium-223 (223Ra) | 1
  None | 1

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Sensitivity of DCFBC-PET as Determined by Agreement of PET/CT Detection of Metastatic Prostate Cancer With Conventional Imaging Modality (CIM)
Description: Measurement of sensitivity of DCFBC PET to CIM (contrast-enhanced CT and bone scintigraphy) for detection of metastatic prostate cancer based on number of lesions that are detected on PET/CT, in agreement with CT and CIM. Measurement of sensitivity were obtained on lesion by lesion analysis where lesions that responded on follow up were considered a true positive.
Time Frame: 24 Months
Population: Combined Imaging Modality (CIM) refers to both CT and BS imaging. The total number of lesions analyzed by both CT and BS (CIM) are 235 (as represented by PET-positive and PET-negative, equivocal CIM). There is overlap in the number of lesions detected by conventional imaging modalities (ie: bone scan and computed tomography)
Measure: Number; unit: lesions detected
Units Other Than Participants: Lesions
Arm/Group | 18F-DCFBC
Number analyzed (Participants) | 17
Number analyzed (Lesions) | 235
lesions detected
  PET Positive, CT negative/equivocal: number analyzed (Lesions) | 170
  PET Positive, CT negative/equivocal | 148
  PET Positive, BS negative/equivocal: number analyzed (Lesions) | 170
  PET Positive, BS negative/equivocal | 170
  PET Positive, Combined CIM negative/equivocal | 170
  PET negative/equivocal, CT positive: number analyzed (Lesions) | 55
  PET negative/equivocal, CT positive | 50
  PET negative/equivocal, BS positive: number analyzed (Lesions) | 55
  PET negative/equivocal, BS positive | 14
  PET negative/equivocal, Combined CIM positive | 55

2. Secondary Outcome: Sensitivity of Detection of New or Progression of Metastasis
Description: Sensitivity of DCFBC-PET and conventional imaging modalities (CIM), which include bone scintigraphy (BS) and contrast-enhanced computed tomography (CECT) to detect new or progression of metastases at follow-up, where "equivocal" lesions are considered negative. Measurement of sensitivity were obtained on lesion by lesion analysis where lesions that responded on follow up were considered a true positive, therefore, sensitivity is a proportion of responsive lesions to the total number of lesions analyzed.
Time Frame: up to 1 year
Population: Follow-up CIM was only available for 12 of the 17 participants. 92% of the lesions detected via 18F-DCFBC PET were marked as true positive.
Measure: Number (95% Confidence Interval); unit: proportion of responsive lesions
Arm/Group | 18F-DCFBC
Number analyzed (Participants) | 12
proportion of responsive lesions
  18F-DCFBC PET | 0.92 [0.80 to 0.97]
  CECT | 0.64 [0.41 to 0.82]
  BS | 0.40 [0.20 to 0.65]
  Combined CIM (BS and CECT) | 0.71 [0.49 to 0.86]

ADVERSE EVENTS:
Time Frame: Up to 1 month
Groups:
- 18F-DCFBC: 18F-DCFBC
Arm/Group | 18F-DCFBC
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 4/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18F-DCFBC (N=17)
Headache (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Blood in stool (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes